CLINICAL TRIAL: NCT04514458
Title: Pragmatic Trial of Messaging to Providers About Treatment of Heart Failure
Acronym: PROMPT-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2000027014
Record Dates: First submitted 2020-07-29; First posted 2020-08-17 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure With Reduced Ejection Fraction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EHR-based alert (Experimental): Providers will receive a best practice alert for each of their eligible patients upon opening of the order entry screen in the patient's medical record. The alert will inform the provider to the presence of HFrEF and of the patient's current left ventricular ejection fraction and current evidence-based medications for HFrEF. It will also provide access to an order set with recommended evidence-based HFrEF therapies as well as a link to the best available guideline-recommended information regarding the treatment of heart failure.
  Interventions: Other: Best practice alert for the notification of patient HFrEF and recommended evidence-based therapies (NO drugs are being administered in this trial)
- Usual Care (No Intervention): Providers will not receive an alert and will proceed with usual care.

INTERVENTIONS:
Other: Best practice alert for the notification of patient HFrEF and recommended evidence-based therapies (NO drugs are being administered in this trial) — Providers will receive a best practice alert for each of their eligible patients upon opening of the order entry screen in the patient's medical record. The alert will inform the provider to the presence of HFrEF and of the patient's current left ventricular ejection fraction and current evidence-based medications for HFrEF. It will also provide access to an order set with recommended evidence-based HFrEF therapies as well as a link to the best available guideline-recommended information regarding the treatment of heart failure.
  Arms: EHR-based alert

SUMMARY:
A randomized controlled trial to compare the efficacy of an electronic health record-based alert informing providers about evidence-based medications for HFrEF versus usual care (no alert) in outpatient clinics across a single health system.

DETAILED DESCRIPTION:
Data from clinical trials suggest that pharmacological therapies prescribed at appropriate doses will lead to dramatic improvements in survival and hospitalization rates in patients with heart failure with reduced ejection fraction (HFrEF). Consequently, major cardiovascular societies assign the highest level of recommendation to use these therapies in all eligible patients. However, data from several registries over the last three decades has failed to see use of these evidence based therapies at levels noted in clinical trials, despite aggressive guideline recommendations and promotion by thought leaders in the field.

It remains unclear as to why many patients with HFrEF are not on evidence-based therapies, and why the percentages are consistent across national registries over time. One explanation might be that providers know the data regarding evidence-based therapies, but the therapies only benefit a narrow population. Another factor might be a lack of knowledge among providers about the appropriate management of HFrEF patients. A simple way to test this hypothesis is to examine whether electronic health record (EHR) based "best practice advisories" (BPAs) can increase use of evidence based therapies. If found to be effective, these low cost interventions can be rapidly applied across large healthcare systems.

This study will conduct a randomized controlled trial across outpatient clinics within a single health system comparing the effectiveness of an EHR-based alerting system that informs practitioners about what evidence-based medications they can prescribe for HFrEF patients versus usual care (no alert). One hundred eligible unique providers will be randomized to an intervention in which an alert will appear for all eligible patients with HFrEF, or to a control group in which no alert appears and usual care will continue, with a target patient enrollment of 1,310. The primary outcome for the trial will be the proportion of patients with HFrEF with an increase in evidence based medical therapies for HFrEF (beta-blockers, ACE-I/ARB/ARNI, MRA, SGLT2i). Secondary outcomes will include 30-day hospital admission rates, 30-day ED visits, one year all-cause mortality, and total 6 month healthcare costs.

ELIGIBILITY:
Patient Inclusion Criteria:

* Age 18 or over
* Seen in eligible internal medicine or cardiology clinic
* Left ventricular ejection fraction less than or equal to 40%
* Registered in the Yale Heart Failure Registry

Patient Exclusion Criteria:

* Opted out of EHR-based research
* Under hospice care
* Already receiving each targeted class of evidence-based HFrEF medical therapy

Selection of Providers:

* Practicing at an eligible internal medicine or cardiology clinic
* High frequency of visits by eligible patients based on retrospective chart review

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1410 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2022-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tariq Ahmad, MD MPH, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Health System selected outpatient clinics, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data underlying results for publication will be made available upon publication of results.
Supporting Information: Study Protocol, SAP
Time Frame: Upon publication of results; indefinitely.

REFERENCES:
- [Derived] Ghazi L, Yamamoto Y, Riello RJ, Coronel-Moreno C, Martin M, O'Connor KD, Simonov M, Huang J, Olufade T, McDermott J, Dhar R, Inzucchi SE, Velazquez EJ, Wilson FP, Desai NR, Ahmad T. Electronic Alerts to Improve Heart Failure Therapy in Outpatient Practice: A Cluster Randomized Trial. J Am Coll Cardiol. 2022 Jun 7;79(22):2203-2213. doi: 10.1016/j.jacc.2022.03.338. Epub 2022 Apr 3. PMID 35385798
- [Derived] Ghazi L, Desai NR, Simonov M, Yamamoto Y, O'Connor KD, Riello RJ, Huang J, Olufade T, McDermott J, Inzucchi SE, Velazquez EJ, Wilson FP, Ahmad T. Rationale and design of a cluster-randomized pragmatic trial aimed at improving use of guideline directed medical therapy in outpatients with heart failure: PRagmatic trial of messaging to providers about treatment of heart failure (PROMPT-HF). Am Heart J. 2022 Feb;244:107-115. doi: 10.1016/j.ahj.2021.11.010. Epub 2021 Nov 20. PMID 34808104

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 100 providers were identified and consented to the study. 93 were randomized to the intervention group (alert) (n=46) or to usual care (no alert) group (n=47). This created 93 clusters (providers) to which eligible patient participants were assigned on their first eligible clinic visit. Eligible patient subjects were automatically identified, enrolled and randomized by our best practice alert based on their provider's randomization status (685 to the intervention group and 625 to usual care).
Pre-assignment Details: 7 provider subjects were excluded prior to randomization as patient recruitment finished before these providers saw an eligible patient.
Period: Overall Study
Arm/Group | EHR-based Alert | Usual Care
Started | 735 | 675
Patient Subjects Enrolled | 685 | 625
Provider Subjects Enrolled | 50 | 50
Completed | 731 | 672
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were not collected for provider subjects. Baseline characteristics are described for patient participants only as the exposure of interest would be expected to affect this study population and primary and secondary outcomes are collected only for patient subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | EHR-based Alert | Usual Care | Total
Number analyzed (Participants) | 685 | 625 | 1310
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 72 [64 to 81] | 72 [62 to 80.8] | 72 [63 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 207 | 195 | 402
  Male | 478 | 430 | 908
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 67 | 58 | 125
  Not Hispanic or Latino | 614 | 559 | 1173
  Unknown or Not Reported | 4 | 8 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 9 | 11 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 119 | 118 | 237
  White | 492 | 447 | 939
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 64 | 48 | 112
Medicaid/Medicare Enrollee [Count of Participants; unit: Participants] | 535 | 582 | 1117
Medical History [Count of Participants; unit: Participants]
  Atrial Arrhythmias | 349 | 342 | 691
  Coronary Artery Disease (CAD) | 262 | 208 | 470
  Chronic Kidney Disease (CKD) | 241 | 212 | 453
  Depression | 124 | 99 | 223
  Diabetes | 260 | 235 | 495
  Dyslipidemia | 524 | 500 | 1024
  Hypertension | 583 | 531 | 1114
  Obesity | 145 | 130 | 275
  Chronic Pulmonary Disorders | 202 | 199 | 401
  Peripheral Vascular Disease | 386 | 392 | 778
Baseline Blood Pressure [Median (Inter-Quartile Range); unit: mmHg]
  Systolic blood pressure | 120 [108 to 130] | 118 [108 to 130] | 120 [108 to 130]
  Diastolic blood pressure | 70 [62 to 78] | 70 [62 to 78] | 70 [62 to 78]
Baseline Heart Rate [Median (Inter-Quartile Range); unit: beats/minute] | 74 [65 to 84] | 74 [65 to 83] | 74 [65 to 84]
Patients per provider type [Count of Participants; unit: Participants]
  Number of patients seen by physician | 467 | 438 | 905
  Number of patients seen by Advanced Practice Providers | 218 | 187 | 405
Number of patients on GDMT classes at baseline [Count of Participants; unit: Participants]
  Beta blockers | 581 | 517 | 1098
  ACE-I/ARB/ARNI | 489 | 437 | 926
  Angiotensin Converting Enzyme Inhibitor (ACE-I) | 93 | 96 | 189
  Angiotensin Receptor Blocker (ARB) | 102 | 91 | 193
  Angiotensin Receptor/Neprilysin Inhibitor (ARNI) | 294 | 250 | 544
  Aldosterone Receptor Antagonist (MRA) | 193 | 186 | 379
  Sodium-Glucose cotransporter-2 inhibitor (SGLT2i) | 83 | 62 | 145
Baseline Potassium [Median (Inter-Quartile Range); unit: mEq/L] | 4.2 [3.9 to 4.6] | 4.3 [4 to 4.68] | 4.3 [4 to 4.6]
Baseline Creatinine [Median (Inter-Quartile Range); unit: mg/dL] | 1.2 [0.95 to 1.6] | 1.2 [0.94 to 1.5] | 1.2 [0.95 to 1.5]
Baseline estimated Glomerular Filtration Rate (eGFR) [Median (Inter-Quartile Range); unit: ml/min/1.73m^2] | 56.9 [40.1 to 76.9] | 58.4 [41.2 to 78.1] | 57.8 [40.7 to 77.5]
Baseline Left Ventricular Ejection Fraction (LVEF) [Median (Inter-Quartile Range); unit: percent ejection fraction] | 32 [24 to 36] | 32 [25 to 37] | 32 [25 to 37]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Heart Failure With Reduced Ejection Fraction (HFrEF) With an Increase in Prescribed HFrEF Therapy
Description: Assessed as an increase in the number of prescribed targeted evidence-based therapies for HFrEF, including beta-blockers, ACEi, ARBs, ARNIs, MRAs, and SGLT2is.
Time Frame: Assessed from the date of randomization to 30 days post-randomization
Population: Observed in patient subjects only.
Measure: Count of Participants; unit: Participants
Arm/Group | EHR-based Alert | Usual Care
Number analyzed (Participants) | 685 | 625
Participants | 176 | 117

2. Secondary Outcome: Percentage of Patients on Beta Blockers
Description: Assessed as the number of patients with prescribed beta blockers
Time Frame: Assessed from the date of randomization to 30 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | EHR-based Alert | Usual Care
Number analyzed (Participants) | 685 | 625
Participants | 606 | 521

3. Secondary Outcome: Percentage of Patients on ACE Inhibitors
Description: Assessed as the number of patients with a prescribed ACEi
Time Frame: Assessed from the date of randomization to 30 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | EHR-based Alert | Usual Care
Number analyzed (Participants) | 685 | 625
Participants | 83 | 92

4. Secondary Outcome: Percentage of Patients on ARBs
Description: Assessed as the number of patients with a prescribed ARB
Time Frame: Assessed from the date of randomization to 30 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | EHR-based Alert | Usual Care
Number analyzed (Participants) | 685 | 625
Participants | 111 | 85

5. Secondary Outcome: Percentage of Patients on ARNIs
Description: Assessed as the number of patients with a prescribed ARNI
Time Frame: Assessed from the date of randomization to 30 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | EHR-based Alert | Usual Care
Number analyzed (Participants) | 685 | 625
Participants | 334 | 285

6. Secondary Outcome: Percentage of Patients on MRAs
Description: Assessed as the number of patients with a prescribed MRA
Time Frame: Assessed from the date of randomization to 30 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | EHR-based Alert | Usual Care
Number analyzed (Participants) | 685 | 625
Participants | 232 | 203

7. Secondary Outcome: Percentage of Patients on SGLT2 Inhibitors
Description: Assessed as the number of patients with a prescribed SGLT2i
Time Frame: Assessed from the date of randomization to 30 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | EHR-based Alert | Usual Care
Number analyzed (Participants) | 685 | 625
Participants | 144 | 103

8. Secondary Outcome: Rate of One-year All-cause Mortality
Description: Assessed as the number of patients who expired from randomization up to one year from any cause.
Time Frame: Assessed from the date of randomization to the date of death from any cause, up to 365 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | EHR-based Alert | Usual Care
Number analyzed (Participants) | 685 | 625
Participants | 75 | 68

9. Secondary Outcome: Rate of 30-day Hospital Admission
Description: Number of participants with a hospitalization within 30 days of randomization
Time Frame: Assessed from the date of randomization to the date of hospital admission, up to 30 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | EHR-based Alert | Usual Care
Number analyzed (Participants) | 685 | 625
Participants | 47 | 63

10. Secondary Outcome: Rate of 30-day All-cause Emergency Department Visits
Description: Number of participants with an emergency department visit within 30 days of randomization.
Time Frame: Assessed from the date of randomization to the date of ED/ER admission, up to 30 days post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | EHR-based Alert | Usual Care
Number analyzed (Participants) | 685 | 625
Participants | 86 | 77

11. Secondary Outcome: Total Six-month Healthcare Costs
Description: Assessed as total direct and indirect cost of patient care from randomization to 6 months post randomization.
Time Frame: Assessed from the date of randomization to 6 months post-randomization
Population: The data necessary to analyze this outcome was unable to be released from the university analytics team, therefore we cannot report cost results. The Finance Administration at Yale did not grant approval for access to this data. The data was not collected and will not be accessed in the future.
Arm/Group | EHR-based Alert | Usual Care
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Percentage of Filled Prescriptions
Description: Proportion of prescriptions filled as assessed by SureScripts
Time Frame: Assessed 6 months post-randomization
Population: Surescripts data is inaccurate and does not capture all patient prescription fills, thus this data cannot currently be obtained.
Arm/Group | EHR-based Alert | Usual Care
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Medication Dose of Any Prescribed Beta Blocker
Time Frame: Assessed at 6 months post-randomization
Population: as for outcome 12
Arm/Group | EHR-based Alert | Usual Care
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Medication Dose of Any Prescribed ACEi
Time Frame: Assessed at 6 months post-randomization
Population: as for outcome 12
Arm/Group | EHR-based Alert | Usual Care
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Medication Dose of Any Prescribed ARB
Time Frame: Assessed at 6 months post-randomization
Population: as for outcome 12
Arm/Group | EHR-based Alert | Usual Care
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Medication Dose of Any Prescribed ARNI
Time Frame: Assessed at 6 months post-randomization
Population: as for outcome 12
Arm/Group | EHR-based Alert | Usual Care
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Medication Dose of Any Prescribed MRA
Time Frame: Assessed at 6 months post-randomization
Population: as for outcome 12
Arm/Group | EHR-based Alert | Usual Care
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Medication Dose of Any Prescribed SGLT2 Inhibitor
Time Frame: Assessed at 6 months post-randomization
Population: as for outcome 12
Arm/Group | EHR-based Alert | Usual Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: One year
Description: Adverse events are reported to the IRB via written report within 5 calendar days of the Principal Investigator becoming aware of the event.
  Adverse events reporting is only described for patient subjects as the exposure of interest would be expected to affect this study population. Adverse events were not monitored or assessed for provider subjects.
Arm/Group | EHR-based Alert | Usual Care
All-Cause Mortality (participants affected / at risk) | 75/685 | 68/625
Serious Adverse Events (participants affected / at risk) | 0/685 | 0/625
Other Adverse Events (participants affected / at risk) | 0/685 | 0/625

LIMITATIONS AND CAVEATS:
Limitations include being conducted at a single health system, that it primarily examined an increase in medication initiation rather than up-titration of dosing, that the alert has only been created and used in the Epic EHR framework, and that the alert was tested during a time when there were coordinated and intensive efforts across the study site to improve medical therapy for heart failure, which is reflected by increases in HFrEF therapies in the usual care arm of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/58/NCT04514458/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/58/NCT04514458/ICF_001.pdf